CLINICAL TRIAL: NCT05255003
Title: STrategies for Anticoagulation in Patients With thRombocytopenia and Cancer-associated Thrombosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tzu-Fei Wang (Other)
Responsible Party: Sponsor-Investigator, Tzu-Fei Wang, Qualified Investigator, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: START Pilot
Record Dates: First submitted 2022-02-06; First posted 2022-02-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cancer-associated Thrombosis; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Enoxaparin; Dalteparin; Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified dose LMWH without platelet transfusion support (Experimental): Patients will be given modified dose LMWH as below based on the first platelet count of the day (daily in admitted patients or at least 2 times a week in outpatients), without empiric platelet transfusion:
  I. Platelet count 25-50,000/µL: 50% dose LMWH
  II. Platelet count < 25,000/µL: hold anticoagulation
  Interventions: Biological: Enoxaparin; Biological: Dalteparin; Biological: Tinzaparin
- Higher dose LMWH with platelet transfusion support (Active Comparator): Patients assigned to higher dose LMWH (see below) will be given transfusion for 14 days when the first platelet count of the day falls below 50,000/uL (daily inpatient or at least 2 times a week in outpatients). Post-transfusion counts will not be routinely obtained unless clinically indicated
  I. Platelet count 25-50,000/µL: platelet transfusion + 100% dose LMWH
  II. Platelet count < 25,000/µL: platelet transfusion + 50% dose LMWH
  After Day 14, patients will be transitioned to modified dose LMWH as the other arm without platelet transfusion.
  LMWH can include enoxaparin, dalteparin, or tinzaparin, with 100% as:
  * Enoxaparin - 1mg/kg subcutaneously twice daily
  * Dalteparin - 200 IU/kg subcutaneously daily for 1 month then 150 U/kg daily
  * Tinzaparin - 175 units/kg subcutaneously daily
  Interventions: Biological: Enoxaparin; Biological: Dalteparin; Biological: Tinzaparin

INTERVENTIONS:
Biological: Enoxaparin — I. Platelet count 25-50,000/µL: 0.5mg/kg subcutaneously twice daily
  II. Platelet count < 25,000/µL: hold anticoagulation
  Other Names: Lovenox
Biological: Dalteparin — I. Platelet count 25-50,000/µL: 100 IU/kg subcutaneously daily for the first month of an acute VTE then 75 U/kg
  II. Platelet count < 25,000/µL: hold anticoagulation
  Other Names: Fragmin
Biological: Tinzaparin — I. Platelet count 25-50,000/µL: 87.5 units/kg subcutaneously daily
  II. Platelet count < 25,000/µL: hold anticoagulation
  Other Names: Innohep

SUMMARY:
Patients with cancer are prone to have blood clots, which are usually treated with blood thinners. The main complication of blood thinners is bleeding. This is especially a concern when the number of platelets in the blood is lower than 50,000 per microliter. The role of platelets is to stop bleeding, so when the number of platelets is low, patients are at a higher risk of bleeding. Cancer patients are prone to have lower platelet numbers due to cancer therapies and/or cancer itself. It is not clear what the best treatment is for cancer patients who need blood thinners for a blood clot but have low platelet counts.

The investigators plan to do a small study called a pilot study to help plan for a larger study in such patients. In the pilot study, investigators will include 50 patients with cancer, low platelet counts, and a blood clot diagnosed within 2 weeks. Patients will be randomly assigned to one of the two treatment strategies: the full dose of blood thinners along with platelet transfusion or a reduced dose of blood thinners without platelet transfusion. The investigators will follow all patients for 30 days. If this pilot study is successful, it will help lead to a much larger trial, which will provide important information on the best treatment strategy for these patients.

DETAILED DESCRIPTION:
The current proposal is for the pilot trial to assess feasibility of a full-scale RCT. To determine feasibility, the pilot and the full-scale trials will use the same recruitment strategy, inclusion/exclusion criteria, interventions, follow up duration, and measurement/adjudication of clinical outcomes. If the pilot trial finds that the full-scale trial is feasible, and no changes to the study design are indicated, the data from the pilot trial will be included in the full-scale trial, which will be efficient and reduce the recruitment time and costs of the full-scale trial.

The START trial is a multi-centre RCT with prospective, open-label, blind-evaluator (PROBE) design. Adult patients with acute cancer-associated thrombosis (diagnosed within 14 days) and thrombocytopenia (platelet count < 50,000/µL) secondary to cancer therapy or cancer itself will be randomized 1:1 to modified dose LMWH or higher dose LMWH with platelet transfusion support, to evaluate the superiority of a modified dose LMWH strategy in reducing clinically relevant bleeding events compared to full dose LMWH with platelet transfusion. The PROBE design is an efficient use of research funds while maintaining the benefits of randomization and blinded evaluation of endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18) with active malignancy (malignancy diagnosed or treated within the previous 6 months, or progressive/relapsed);
2. Objectively confirmed VTE within last 14 days for which therapeutic anticoagulation is planned;
3. Thrombocytopenia with a platelet count < 50,000/uL from cancer therapy or malignancy itself;
4. Able to provide written informed consent

Exclusion Criteria:

1. Receipt of anticoagulant for index VTE with platelet count < 50,000/uL for > 72 hours;
2. Superficial vein thrombosis only;
3. Life expectancy < 1 month (as judged by the treating physicians);
4. Creatinine clearance < 30 ml/min;
5. Contraindication to LMWH such as a history of heparin induced thrombocytopenia;
6. Thrombocytopenia from other causes, such as thrombotic microangiopathy, immune thrombocytopenia, disseminated intravascular coagulation;
7. Previously documented history of refractoriness to platelet transfusion secondary to HLA antibodies;
8. Refusal of blood products;
9. Anticoagulation at any dose is deemed unsafe (i.e. active bleeding or bleeding disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - The average number of patients recruited per month | 18 months
  The average number of patients recruited per month

SECONDARY OUTCOMES:
Feasibility - Proportion of eligible patients who provide consent | 18 months
  Number of consenting participants from the number of eligible patients
Feasibility - Reasons for non-participation in eligible patients | 18 months
  Reasons for non-participation in eligible patients
Feasibility - Number of patients who complete study procedures by adhering to protocol | 18 months
  Number of participants adhering to the protocol (such as anticoagulation, transfusion, platelet count monitoring according to the protocol)
Feasibility - Rates of withdrawal | 18 months
  Number of participants withdrawing from study
Feasibility - Loss to follow-up | 18 months
  Number of participants lost to follow-up
Feasibility - Crossover between treatment arms | 18 months
  Number of participants crossing over between treatment arms
Clinical Outcome - Rate of clinically relevant bleeding (composite of major bleeding and clinically relevant non-major bleeding events) | 18 months
  Rate of clinically relevant bleeding (composite of major bleeding and clinically relevant non-major bleeding events)
Clinical Outcome - Rate of symptomatic or incidentally detected recurrent or new major VTE | 18 months
  Rate of symptomatic or incidentally detected recurrent or new major VTE
Clinical Outcome - PE-related death | 18 months
  PE-related death
Clinical Outcome - Composite of recurrent VTE and major bleeding events | 18 months
  Composite of recurrent VTE and major bleeding events
Clinical Outcome - Non-major VTE (distal upper or lower extremity DVT, superficial upper or lower extremity vein thrombosis) | 18 months
  Number of non-major VTE (distal upper or lower extremity DVT, superficial upper or lower extremity vein thrombosis)
Clinical Outcome - Duration of thrombocytopenia (days of platelet count < 50,000/uL) per patient | 18 months
  Duration of thrombocytopenia (days of platelet count < 50,000/uL) per patient
Clinical Outcome - Number of transfused units and adverse platelet transfusion reactions | 18 months
  Number of transfused units and adverse platelet transfusion reactions
Clinical Outcome - Overall mortality | 18 months
  Overall mortality
Clinical Outcome - Health-related quality of life using EuroQoL-EQ-5D-5L questionnaire | 18 months
  Health-related quality of life using EuroQoL-EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Fei Wang, MD, Principal Investigator — Ottawa Hospital Research Institute; Marc Carrier, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health - St. Catharines Site, Saint Catharines, Ontario
  - Windsor Regional Hospital, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No